CLINICAL TRIAL: NCT02438215
Title: An Open-Label, Single Site Study Using [123I]β-CIT Single Photon Emission Tomography (SPECT) to Evaluate Dopamine Transporter Binding Following Treatment With IRX4204 in Early Parkinson's Disease Subjects
Brief Title: Study of IRX4204 for Treatment of Early Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Io Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRX4204-001
Record Dates: First submitted 2014-08-07; First posted 2015-05-08 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's Disease
Keywords: PD; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — IRX4204; AGN 194204

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IRX4204 (Experimental): IRX4204 20 mg QD for Days 1-30
  Interventions: Drug: IRX4204

INTERVENTIONS:
Drug: IRX4204 — IRX4204 is a potent and highly selective orally available and brain penetrant RXR nuclear receptor agonist small compound administered as gel capsules.
  Other Names: NRX194204

SUMMARY:
This is a single site, open-label study designed to examine dopamine transporter density using [123I]β-CIT SPECT imaging before and following treatment with IRX4204 for a 30-day period in early Parkinson's disease patients. In addition, clinical evaluations will be performed to evaluate the effect of IRX4204 treatment on the motor and cognitive symptoms of PD.

DETAILED DESCRIPTION:
Fifteen patients with early PD were enrolled in this open label study, in 3 cohorts of 5 patients each, treated with IRX4204 at 5 mg/day, 10mg/day, or 20 mg/day. Patients were administered IRX4204 orally once daily. Baseline assessments were performed for total motor score, and Unified Parkinson's Disease Rating Scale (UPDRS). Follow-up assessments of these clinical outcome measures were performed at 14 and 29 days of treatment. [123]β-CIT SPECT imaging for assessment of dopamine active transporter (DAT) expression was performed at baseline, and on day 30 of IRX4204 treatment. Patients had clinical hematology and chemistry laboratory tests, and recording of adverse events, performed at baseline and at follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 40-80 years of age, inclusive.
2. Participant has a clinical diagnosis of PD based on the UK Brain Bank Criteria.
3. Participant has Hoehn and Yahr stage < 3.
4. Participant may be treated with PD symptomatic therapy on a stable dose for at least 30 days prior to the Screening Visit. Dose levels of PD symptomatic therapies will remain stable through the patient's participation in the study, unless a change of dose level is indicated because of adverse events.
5. Participant must be willing and able to provide informed consent.
6. Females must be of either non-child bearing potential based on:

   * post-menopausal for at least 2 years, or
   * surgically sterilized If of child bearing potential, must be neither pregnant or breastfeeding at Screening, and must be willing to avoid pregnancy by using medically accepted contraception (use of an intrauterine device or use of a double barrier method when engaging in sexual intercourse with a male partner) for 4 weeks prior to and 4 weeks following the last dose of study medication.

Exclusion Criteria:

1. Has any form of parkinsonism other than idiopathic PD
2. Are currently experiencing motor fluctuations (end of dose wearing off or dyskinesias) reflective of later stage PD
3. Has evidence of dementia or significant cognitive dysfunction
4. Has clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
5. The subject has any disorder that may interfere with drug absorption, distribution, metabolism or excretion.
6. The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
7. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
striatal binding ratio (SBR) | 30 days
  The percent change from baseline to end of dosing period (Day 30) of the striatal binding ratio (SBR)

SECONDARY OUTCOMES:
Total Motor and UPDRS scores | 30 days
  The change in motor and UPDRS scores to end of dosing period (Day 30)
Safety including hematology and chemistry laboratories, vital signs, and adverse events | 30 Days
  Clinically significant changes in hematology and chemistry laboratories, vital signs, and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ken Marek, MD, Principal Investigator — Molecular NeuroImaging, [MNI]
Locations (1):
- Molecular NeuroImaging, [MNI], New Haven, Connecticut, United States